CLINICAL TRIAL: NCT05647733
Title: Effects of an Intraoperative Low-splanchnic Blood Volume Restrictive Fluid Management Strategy Compared to a Cardiac Output Optimized Liberal Fluid Management Strategy on Postoperative Outcomes in Liver Transplantation
Brief Title: Restrictive Fluid Management In Liver Transplantation (REFIL)
Acronym: REFIL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Donation and Transplantation Research Program (CDTRP) (Unknown); Canadian Perioperative Anesthesia Clinical Trial (PACT) Group (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2023-11173
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Liver Transplantation
Keywords: Hemodynamic management; Fluid management; Transfusions; Phlebotomy
MeSH Terms: interventions — Phlebotomy

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to either group in a 1:1 ratio. A research assistant will randomize the patient once a viable graft is confirmed, and then share allocation with the anesthesiology team.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Only the anesthesiology team will know the allocation received since they must implement the intervention, limiting differential outcome classification bias since they will not assess outcomes. Patients, surgeons, and non-anesthesia health professionals will be blinded to allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restrictive group: Low splanchnic blood volume Restrictive fluid management strategy (Experimental): The intervention group is targeted at lowering splanchnic blood volume using a phlebotomy and restricting fluid infusion, individualized to the physiological needs of this population and the distinct LT surgical phases. The strategy will first consist of performing a phlebotomy without fluid replacement at the start of surgery.We will combine it with fluid restriction to prevent excessive fluid administration and its effect on splanchnic blood volume and blood loss, combined with the effect of the phlebotomy, as well as to limit fluid overload, as previously reported. Fluid will be administered to compensate blood loss and treat severe hemodynamic instability.The phlebotomy will be transfused back at the beginning of the reperfusion phase where fluid management will be based on a goal-directed therapy (GDT) using either PPV or SV, as in the control group.
  Interventions: Procedure: Low splanchnic blood volume restrictive fluid management strategy; Procedure: Phlebotomy
- Liberal group: Optimized cardiac output liberal fluid management strategy (Active Comparator): The control group will receive a liberal intraoperative fluid management strategy optimizing cardiac output throughout the surgery. It will consist of administering 250 mL fluid boluses until SV stops to increase by more than 10% or until PPV is below 12%, a dynamic indicator of fluid responsiveness validated in many surgical populations, including ESLD patients undergoing a LT.This strategy is informed by data from recent clinical trials on benefits of GDT in major surgery, data on strategies used in major surgery, liver resection or LT and our survey on current practice.
  Interventions: Procedure: Optimized cardiac output liberal fluid management strategy

INTERVENTIONS:
Procedure: Low splanchnic blood volume restrictive fluid management strategy — Hemodynamic goal-directed restrictive fluid management strategy.
  Other Names: Restrictive arm
  Arms: Restrictive group: Low splanchnic blood volume Restrictive fluid management strategy
Procedure: Optimized cardiac output liberal fluid management strategy — Permissive intraoperative hemodynamic goal-directed fluid management strategy that optimizes cardiac output throughout surgery
  Other Names: Liberal arm
  Arms: Liberal group: Optimized cardiac output liberal fluid management strategy
Procedure: Phlebotomy — Retrieval of blood in a blood donation bag performed prior to dissection and transfused back after graft reperfusion
  Arms: Restrictive group: Low splanchnic blood volume Restrictive fluid management strategy

SUMMARY:
Hypothesis: A Canadian multicentre clinical trial is feasible. Study Design: Multicenter internal pilot parallel arm randomized controlled trial

Study population: Patients with end-stage liver disease undergoing a liver transplantation not meeting any exclusion criteria.

Primary endpoint: The primary feasibility endpoint is an overall recruitment rate ≥ 4 patients/month across all three participating sites.

Secondary endpoint: The secondary feasibility endpoints are a protocol adherence > 90%, a 30-day (or hospital discharge) and 6-month outcome measurement > 90%, and a mean difference in total intraoperative volume received (crystalloids and colloids combined) > 1000 ml between groups.

Study intervention: Low splanchnic blood volume restrictive fluid management strategy (intervention). A phlebotomy, performed prior to dissection and transfused back after graft reperfusion, combined with a hemodynamic goal-directed restrictive fluid management strategy

Optimized cardiac-output liberal fluid management strategy (control) A hemodynamic goal-directed liberal fluid management strategy that optimizes cardiac output throughout surgery

DETAILED DESCRIPTION:
MAIN OBJECTIVE The main objective of the REFIL-1 pilot study is to establish the feasibility (recruitment, adherence, outcome measurement) of conducting a Canadian multicentre randomized controlled trial comparing an intraoperative low-splanchnic blood volume restrictive fluid management strategy to a cardiac output optimised liberal fluid management strategy in adult LT for ESLD. The hypothesis is that a Canadian multicentre clinical trial is feasible.

SECONDARY OBJECTIVES The overarching objective of the ReFIL (Restrictive Fluid management In Liver transplantation) research program, which will be answered in a future large-scale trial, regards the efficacy of the proposed interventional strategy to improve postoperative outcomes in LT.

TERTIARY OBJECTIVES Our tertiary objective is to measure the cost-effectiveness of the proposed intervention based on the composite outcome of any severe postoperative complications and graft loss.

DESIGN AND STUDY POPULATION This study a multicentre internal pilot parallel arm randomized trial comparing two intraoperative hemodynamic and splanchnic blood volume management strategies in LT recipients.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient ≥ 18 years of age undergoing liver transplantation for ESLD.

Exclusion Criteria:

* Patients undergoing LT for an indication other than ESLD such as acute liver failure, liver cancer without ESLD, retransplantation, amyloid neuropathy or any other indication not associated with ESLD.
* Patients undergoing a combined liver and lung or liver and heart transplantation.
* Patients with any of the following conditions:
* severe chronic renal failure (GFR < 15 ml/minute/1.73 m2 [CKD-EPI equation] or already on RRT);
* severe anemia (hemoglobin level < 80 g/L);76,93,109
* hemodynamic instability (norepinephrine equivalent > 10 ug/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-04-25 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 18 months (at study level)
  Overall recruitment rate ≥ 4 patients/month (across all sites)
Adherence | At time of surgery
  Protocol adherence > 90%, defined using a questionnaire
Hospital outcome measurement completeness | At 30 days (or hospital discharge) after surgery
  A 30 days or hospital discharge outcome measurement > 90%
6-month outcome measurement completeness | 6 months after surgery
  6-month outcome measurement > 90%
Mean difference in total volume received | At time of surgery
  A mean difference in total volume received (crystalloids and colloids combined) > 1000 ml between groups.

SECONDARY OUTCOMES:
Severe complications and graft lost | Up to 30 days or hospital discharge
  Composite incidence of severe complication (Dindo-Clavien III or more) or graft lost (retransplantation or death)
Intraoperative blood loss | End of surgery
  Intraoperative blood loss in mL
Intraoperative and perioperative blood product transfusions | From randomization up to 30 days or hospital discharge, whichever comes first
  Total number of transfused units of labile and non-labile blood products (red blood cells, plasma, platelets, cryoprecipitates, fibrinogen, prothrombin complex concentrates)
7-day quality of recovery | 7 days after surgery
  7-day quality of recovery measured using the QoR-15 (Quality of Recovery) tool
7-day graft dysfunction | 7 days after surgery
  7-day graft dysfunction (definition as reported by Olthoff et al.)
7-day AKI (grade 2 or 3) | 7 days after surgery
  7-day AKI grade 2 or 3 using the KDIGO (Kidney Disease: Improving Global Outcomes) definition
Any complication | From randomization up to 30 days or hospital discharge, whichever comes first
  Any of the following complications, graded according to the Dindo-Clavien classification system: hemorrhagic, graft related, pulmonary, infectious or thromboembolic.
Any other severe complication | From randomization up to 30 days or hospital discharge, whichever comes first
  Any other severe complication (Dindo-Clavien III or more)
Organ dysfunction and support | 30 days
  30-day organ support free days, using a recognized definition (as reported by Heyland et al.)
Intensive care unit (ICU) length of stay | From randomization up to hospital discharge (ascertained up to end of follow-up at 1 year)
  Total duration of stay (days) in the intensive care unit (ICU)
Hospital length of stay | From randomization up to hospital discharge (ascertained up to end of follow-up at 1 year)
  Total duration of stay (days) in the hospital
Quality of life (QoL) | 6 & 12 months after surgery
  Quality of life (QoL) using the SF-36 tool
Hospital readmissions | From randomization up to 1 year after surgery
  Hospital readmissions
Graft complications | From randomization up to 1 year after surgery
  Graft complications
Survival | From randomization up to 1 year after surgery
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Francois-Martin Carrier, MD, Principal Investigator — Centre hospitalier université de Montréal
Locations (3):
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No
End-of-grant KT modalities will be used to reach other important stakeholders, researchers and members of the anesthesia and transplantation community: scientific meetings, publication in an open-access journal, and public presentations with patient partners. Knowledge diffusion on potential difficulties of conducting such trials (and solutions) will be transferred to the research community through the Canadian Perioperative Anesthesia Clinical Trial group (PACT), the Canadian Donation and Transplantation Research Program (CDTRP) and the International Liver Transplantation Society (ILTS) meetings.